CLINICAL TRIAL: NCT01878643
Title: Pilot Study of the Effects of Inhaled Antibiotic on Bacterial Resistance
Brief Title: Reduction of Bacterial Resistance With Inhaled Antibiotics in the Intensive Care Unit
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20033799
Record Dates: First submitted 2013-06-07; First posted 2013-06-17 (Estimated); Last update posted 2013-06-17 (Estimated); Status verified 2013-06

CONDITIONS: Respiratory Infection; Bacterial Resistance; Respiratory Failure
Keywords: aerosolized antibiotic; ventilator-associated pneumonia; bacterial resistance; ventilator -associated tracheobronchitis; clinical pulmonary infection score
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Insufficiency; Pneumonia, Ventilator-Associated | interventions — Vancomycin; Gentamicins; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drug: Placebo (Placebo Comparator): normal saline 2 mL nebulized Q 8 hours placebo for gentamicin or vancomycin
  Interventions: Drug: Placebo
- Drug: vancomycin or gentamicin (Experimental): vancomycin 120 mg every 8 hours or gentamicin 80 mg every 8 hours
  Interventions: Drug: vancomycin or gentamicin

INTERVENTIONS:
Drug: vancomycin or gentamicin — Choice of antibiotic is determined by Gram stain of sputum.The antibiotic is administered via nebulization through the ventilator circuit every 8 hours
  Other Names: gentamicin sulfate; vancomycin hydrocloride
  Arms: Drug: vancomycin or gentamicin
Drug: Placebo — normal saline administered to patient via nebulization
  Other Names: Normal saline 2mL
  Arms: Drug: Placebo

SUMMARY:
The purpose of this study was :

* to determine the effect of inhaled antibiotics on airway bacteria in ventilated patients
* to determine the effect of inhaled antibiotics on respiratory infection

DETAILED DESCRIPTION:
Double-blind randomized placebo controlled study examining the effect of aerosolized antibiotics on respiratory infection signs and symptoms and on bacterial eradication and resistance.

Systemic antibiotics are administered by the responsible physician

ELIGIBILITY:
Inclusion Criteria:

* be on mechanical ventilation greater than 3 days
* greater than or equal to 18 years and survival greater than 14 days
* organisms on Gram stain with increasing purulent secretions

Exclusion Criteria:

* pregnancy
* allergy to drugs administered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2001-12; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

PRIMARY OUTCOMES:
Eradication of multi-drug resistant bacteria | Randomization and at end of treatment
  Tracheal aspirates are taken at randomization. Randomization to drug is determined by the Gram stain(organisms are Gram-positive, Gram-negative or both). End of treatment culture, susceptibility and Gram stain of tracheal aspirate is taken after 14 days of treatment or at time of extubation, (which ever comes first).
  Eradication is defined as absence of growth in culture and absence of organisms on Gram stain.

SECONDARY OUTCOMES:
Clinical Pulmonary Infection Score (CPIS) | Randomization and at end of treatment which is defined as 14 days or at time of extubation, which ever comes first.
  CPIS is an index for risk of respiratory infection using a number of signs and symptoms . An index of greater than or equal to 6 suggests pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Lucy B Palmer, MD, Principal Investigator — Stony Brook University
Locations (1):
- University Hospital Medical Center, Stony Brook, New York, United States

REFERENCES:
- [Derived] Palmer LB, Smaldone GC. Reduction of bacterial resistance with inhaled antibiotics in the intensive care unit. Am J Respir Crit Care Med. 2014 May 15;189(10):1225-33. doi: 10.1164/rccm.201312-2161OC. PMID 24646034